CLINICAL TRIAL: NCT02900365
Title: Early Vs Late Post Traumatic Cataract Surgery and Intraocular Lens Implantation
Brief Title: Early Vs Late Post Traumatic Cataract Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Farabi Eye Hospital (Other)
Responsible Party: Principal Investigator, mohammad soleimani, Assistant Professor, Farabi Eye Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 17865
Record Dates: First submitted 2016-03-27; First posted 2016-09-14 (Estimated); Last update posted 2016-09-14 (Estimated); Status verified 2016-09

CONDITIONS: Traumatic Cataract
Keywords: trauma; cataract; lensectomy; time; early; late
MeSH Terms: conditions — Wounds and Injuries; Cataract

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Early cataract surgery group (Experimental): Eyes which presented with cataract and underwent surgery within 1 week were included in the early procedure group. They underwent "early cataract surgery & IOL implantation"
  Interventions: Procedure: early cataract surgery & IOL implantation
- Late cataract surgery group (Experimental): Eyes which presented with cataract and underwent surgery at least 1 month after trauma were included in the secondary procedure group.They underwent "Late cataract surgery & IOL implantation".
  Interventions: Procedure: late cataract surgery & IOL implantation

INTERVENTIONS:
Procedure: early cataract surgery & IOL implantation — first week cataract extraction and IOL implantation.
  Arms: Early cataract surgery group
Procedure: late cataract surgery & IOL implantation — first month cataract extraction and IOL implantation.
  Arms: Late cataract surgery group

SUMMARY:
In a randomized clinical trial, 30 eyes with traumatic cataract after open globe injury with IOL implantation underwent early and 30 eyes underwent late cataract surgery. We excluded patients who were under 12-year-old. All patients were visited at 1week, 4 weeks , 12 weeks and six months after surgery. In each visit, patients were examined regarding visual acuity, intraocular pressure (IOP), anterior chamber inflammation, IOL position and posterior synechiae. In addition, posterior segment evaluation and funduscopy were performed. Intraoperative complication including posterior capsular rupture, anterior vitrectomy and zonulysis as well as the site of IOL implantation were documented and postoperative complications including raised IOP, anterior chamber inflammation, visual axis opacity, posterior synechiae, subluxation of IOL, IOL pigment deposition were listed.

DETAILED DESCRIPTION:
In a randomized clinical trial, 30 eyes with traumatic cataract after open globe injury underwent early (during the first week after the trauma) (Group 1) and 30 eyes underwent late cataract surgery (after one month of the trauma) (Group 2) (Figure 1a). All cases were observed for at least a 6-month period after the surgery.

Inclusion criteria included patients older than 12-year-old with significant traumatic cataract after open globe injury. Exclusion criteria included patients with anterior capsule rupture as well as disseminated lens materials in the anterior chamber (Figure 1b), patients with hypopyon, eyes undergoing simultaneous primary repair and cataract extraction, cases that IOL implantation was not possible and patients with direct trauma to the posterior segment or with lacerations associated with vitreous prolapse.

In those cases, that IOL power calculation was not possible by the biometry of the affected eye, it was performed using the biometry of the fellow eye. The Ethics Committee of Tehran University of Medical Sciences approved the conduction of the present study and all procedures started after written informed consent was obtained following the explaining the possible consequences of the different methods of treatment to patients. All procedures were performed by the same surgeon (M.B.R.).

All cases underwent lensectomy using vitrectomy probe through the limbal incision. We excluded those patients who needed pars plana vitrectomy from the study. Anterior capsulectomy was performed using a vitrectomy probe and anterior vitrectomy was performed in cases of posterior capsular rupture or vitreous prolapse because of zonular dehiscence. If there was a too hard nuclear part for the vitrectomy probe, we emulsified and suctioned the nucleus using a phacoemulsification handpiece. If the capsular integrity permitted, a posterior chamber IOL was implanted. In this situation, if posterior capsule was not intact, a three piece acrylic foldable (Alcon MA60) IOL was implanted. In other situations, a one-piece foldable acrylic (Alcon SA60) IOL was implanted.

Patients were randomly assigned for early or late cataract extraction and IOL implantation. Randomization was based on a computer-generated sequence based on permuted block randomization method. The length of blocks varied randomly between two, four and six patients. A biostatistician performed the randomization and the sequence of randomization was concealed from the investigators.

All patients received prophylactic oral antibiotic therapy (ciprofloxacin 750 mg twice daily for three days) following the open globe injury. (1). Following surgery, topical antibiotics, corticosteroids and cycloplegics were prescribed and then topical steroids were continued for four weeks and tapered gradually during this period.

We visited all patients at 1week, 4weeks and 12 weeks and 6 months after surgery. In each visit, patients were examined regarding visual acuity, intraocular pressure (IOP), anterior chamber inflammation, IOL position and posterior synechiae. In addition, posterior segment evaluation and funduscopy were performed. Anterior chamber inflammation assessed by Standardization of Uveitis Nomenclature (SUN) Working Group grading scheme for anterior chamber cells and flare and grade ≥2+ was considered significant (14). BCVA ( best corrected contact lens visual acuity) of both eyes was evaluated in logMAR at six months of follow up visits. Another surgeon who did not know timing of the surgery (M.S.) performed this evaluation.

Sample size was calculated as 30 eyes to have a power of 90% to detect a difference of 0.2 logMAR in BCVA between the two groups when the standard deviation of BCVA was assumed to be 0.24 logMAR and the type I error was 0.05 for two-sided test. To assess for the normal distribution of data we used Q-Q plot and Kolmogorov-Smirnov test. To describe data we used mean, standard deviation, median and range. To compare the results between two groups we used t-test, Mann-Whitney, Fisher exact and Chi-Square tests. All statistical methods were performed using SPSS software (IBM Corp. Released 2013. IBM SPSS Statistics for Windows, Version 22.0. Armonk, NY: IBM Corp.). P-values less than 0.05 were considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Eyes which presented with cataract and underwent surgery within 1 week were included in the early procedure group.
* Eyes which presented with cataract and underwent surgery at least 1 month after trauma were included in the secondary procedure group.

Exclusion Criteria:

* Eyes that primary repair and cataract extraction were done at the same time excluded from the study (because these eyes had anterior capsular rupture and disseminated lens material in the anterior chamber necessitating early surgery).
* Also cases that IOL implantation was not possible at the time of cataract extraction were excluded.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-03; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
BCVA | 6 months
  best corrected visual acuity

SECONDARY OUTCOMES:
Posterior capsular rupture | during operation
  Posterior capsular rupture during operation
inflammation | 6 month
  Anterior chamber inflammation assessed by Standardization of Uveitis Nomenclature (SUN) Working Group grading scheme for anterior chamber cells and flare and grade ≥2+ was considered significant

IPD SHARING:
Plan to Share IPD: No